CLINICAL TRIAL: NCT03110484
Title: SAMSUNG MEDICAL CENTER
Brief Title: Pemetrexed in Combination With Erlotinib as a Salvage Treatment in Patients With Metastatic Biliary Tract Cancer (BTC) Who Failed Gemcitabine Containing Chemotherapy: A Phase II Single Arm Prospective Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Seung tae Kim,PhMD, Samsung Medical Center, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-06-111
Record Dates: First submitted 2017-04-07; First posted 2017-04-12 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Pemetrexed; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pemetrexed+Tarceva (Experimental): D1 Pemetrexed 500 mg/m2 IV+ D1-21 Erlotinib 100mg once daily
  Interventions: Drug: Pemetrexed 500 MG; Drug: Erlotinib

INTERVENTIONS:
Drug: Pemetrexed 500 MG — Pemetrexed 500 mg/m2
Drug: Erlotinib — Erlotinib 100mg once daily

SUMMARY:
Pemetrexed in combination with erlotinib as a salvage treatment in patients with metastatic biliary tract cancer (BTC) who failed gemcitabine containing chemotherapy

DETAILED DESCRIPTION:
Biliary tract carcinoma (BTC) is rare in the Europe and the United States, but not uncommon in Asia and Latin America. The tumor arises from the ductular epithelium of the biliary tree within the liver (intrahepatic), the extrahepatic ducts (extrahepatic), or the gallbladder. Intrahepatic cancer is steadily increasing in the Western world. BTCs carry a poor prognosis with 1-year survival rate of 25%. Although surgery remains the only curative treatment for BTC, most patients present with advanced disease and die within a few months of diagnosis. While a combination of gemcitabine and platinum agents seems to be a conclusive treatment option as first-line treatment until now, the role or the optimal regimen for second-line treatment has not been established.

Pemetrexed, a multitarget antifolate which inhibits thymidylate synthase, dihydrofolate reductase and glycinamide ribonucleotide formyltransferase, was approved for the treatment of lung cancer and mesothelioma. In addition to its therapeutic efficacy, pemetrexed has tolerable safety profile and is considered as important therapeutic option for patients of poor performance statue or older age. Pemetrexed was studied in combination with gemcitabine in BTC patients and needs further research in BTC patients. Erlotinib is EGFR tyrosine kinase inhibitor. In BTC and pancreatic cancer, erlotinib showed prolonged survival in combination with chemotherapy. Moreover, the addition of erlotinib to gemcitabine and oxaliplatin showed antitumour activity in our previous phase III trial. And combination of pemetrexed and erlotinib showed tolerable safety profile in lung cancer trial.

So we plan this study to evaluate the efficacy and safety of pemetrexed in combination with erlotinib as a second line treatment in biliary tract cancer

ELIGIBILITY:
Inclusion Criteria:

Provision of a signed written informed consent Age ≥ 20 Histologically or cytologically confirmed carcinoma of biliary tract (intrahepatic, extrahepatic cholangiocarcinoma and gall bladder cancer) Unresectable or metastatic Progression after treatment with first line gemcitabine-based chemotherapy ECOG performance status of 0~2 Measurable lesion per RECIST 1.1 criteria Expected life expectancy ≥ 3months Adequate marrow, hepatic, renal and cardiac functions

Exclusion Criteria:

Poor performance statue Other primary cancer except properly treated non-melanoma skin cancer, cured cervix carcinoma in situ and other cured solid tumor without evidence of recurrence after 5 years of curative treatment.

Severe co-morbid illness and/or active infections Any other clinical trial therapeutics within 14 days Any anti-cancer therapy within 3 weeks prior to initiation of study treatment (radiotherapy, systemic chemotherapy) CTCAE grade 2 or more adverse events remained except alopecia QTcB > 480msec or family history of QT prolongation Current heart problem such as: pooly controlled hypertension

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-07-09 (Actual); Primary Completion 2023-06-14 (Estimated); Study Completion 2024-06-14 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 18MONTHS
  Overall response rate

CONTACTS AND LOCATIONS:
Overall Officials: seungtea kim, Principal Investigator — SamsungMedicalCenter
Locations (1):
- Samsung Medical Center, Seoul, South Korea